CLINICAL TRIAL: NCT03144037
Title: Adherence of Hispanic / Latina Breast Cancer - Patients to Adjuvant Aromatase Inhibitors - (AIs)
Brief Title: Adherence of Hispanic / Latina Breast Cancer - Patients to Adjuvant Aromatase Inhibitors
Acronym: ALPA
Status: Completed | Type: Observational
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Alexander Philipovskiy, Assistant Professor, Texas Tech University Health Sciences Center, El Paso
Other Study IDs: E17086
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational trial designed to assess prospectively the adherence rate to AIs among women with invasive breast cancer (stages I-III) currently receiving AI adjuvant therapy after standard local and systemic therapy. We will study adherence by administrating the 8-item Morisky Medication Adherence Scale (MMAS - 8).

DETAILED DESCRIPTION:
* Women with breast cancer seen at the Texas Tech Physicians Breast Care Center will be recruited during their routine follow-up visit with their medical oncologist.
* Post - menopausal women with histologically confirmed hormonal positive (ER and/or PR) invasive breast cancer stages I - III with no evidence of metastatic disease (M0).
* Patients must be on one of AI (steroidal or non-steroidal).
* Patient must have completed local treatment (surgery /radiation) and recovered from all side effects of chemotherapy and surgery.
* Patient must be able to complete a demographic and the MMAS - 8 questionnaires in English or Spanish.

ELIGIBILITY:
Inclusion Criteria:

* Post - menopausal women with histologically confirmed hormonal positive (ER and/or PR) invasive breast cancer stages I - III with no evidence of metastatic disease (M0).
* Patient must have completed local treatment (surgery /radiation) and recovered from all side effects of chemotherapy and surgery.
* Patient must be on one of AI (steroidal or non-steroidal).
* Patient must be able to complete a demographic and the MMAS - 8 questionnaires in English or Spanish

Exclusion Criteria:

* < 18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Majority of patients are females who are currently on AIs.
Study Population: Hispanic population is targeted, yet study is open for all those who qualify.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Adherence rate per the 8-item Morisky Medication Adherence Scale (MMAS - 8). | Every 6 months for up to 24 months
  Primary endpoint of this study is to determine the adherence rate (high, medium and low) through the MMAS-8 among early stage breast cancer patients being treated at Texas Tech University Health Sciences Center El Paso (TTUHSC EP) where the majority of the patients are of Hispanic origin.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Philipovskiy, MD, PhD, Principal Investigator — Texas Tech University Health Sciences Center, El Paso
Locations (1):
- Texas Tech University HSC El Paso, El Paso, Texas, United States